CLINICAL TRIAL: NCT01591642
Title: Physical Activity, Functional Fitness and Quality of Life After Coronary Artery Bypass Grafting
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FEMH-IRB-099087-E
Record Dates: First submitted 2012-04-27; First posted 2012-05-04 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2010-10

CONDITIONS: Coronary Artery Bypass Graft
Keywords: physical activity; functional fitness; quality of life
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The main purposes of this study are: (1) to investigate the difference of the physical fitness, and quality of life (QOL) among different physical activity levels in post-coronary artery bypass graft (CABG) patients; (2) to analyze the relationships between physical activity and physical fitness and QOL in this population. The investigators predict physical activity and physical fitness remain limited in patients after CABG, and patients with higher physical activity levels will have higher QOL and physical fitness.

DETAILED DESCRIPTION:
Heart diseases continue as the top 3 causes of death in Taiwan in recent ten years. Coronary artery disease (CAD) is the most prevalent fatal heart disease. Coronary artery bypass graft surgery (CABG) is now one of the most common procedures to treat CAD. It was reported that CABG intervention could prolong the life. However, outcomes of CABG have historically been measured in terms of mortality and recurrence of symptoms or complications.There is ample evidence to demonstrate the effect and benefit of cardiac rehabilitation in QOL and function activity in patients post CABG. However, the participation rate of postoperative cardiac rehabilitation is low, especially in women.Little research has been done to examine the physical activity, physical performance, and QOL in this population outside the cardiac rehabilitation setting.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing CABG without valve surgery

Exclusion Criteria:

1. systemic disease, such as liver, renal disease,
2. amputation,
3. cerebrovascular disease or any others disease with limbs dysfunction,
4. lung deficit,
5. cancer,
6. cognitive disorders.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: . All patients who underwent CABG at the Department of Cardiovascular Center at Far-Eastern Memorial Hospital since January 2000 were selected for recruitment to this study.
Sampling Method: Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
physical activity | The participants were followed at one time points after operation in past 10 years
  The level of physical activity was evaluated by the self-administrated long form of the International Physical Activity Questionnaire, which was permitted by the Bureau of Health Promotion, Department of Health, R.O.C.(Taiwan). It is an instrument that estimates the weekly time spent on the performance of physical activities according to intensity, in different contexts of life (workplace, household tasks, transport and leisure). Reported minutes per week in each category were weighted by a metabolic equivalent (MET; multiples of resting energy expenditure).

SECONDARY OUTCOMES:
physical fitness | The participants were followed at one time points after operation in past 10 years
  Physical fitness The outcome measures of physical fitness included body mass index(BMI), waist circumference(WC), grip strength, 30-second chair stand test, and six-minute walk test(6MWT).
quality of life | The participants were followed at one time points after operation in past 10 years
  QOL was measured using abbreviated version of the World Health Organization Quality of Life (WHOQOL-BREF) questionnaire. The original WHOQOL-BREF comprised 26 questions and included four domains: physical, psychological, social relationships, and environment. The WHOQOL-BREF scale has been adapted for Taiwan and added two questions appropriate for Taiwanese culture.